CLINICAL TRIAL: NCT03297879
Title: Beijing Chao-Yang Hospital, Capital Medical University
Brief Title: Comparison of Exenatide and Metformin Monotherapy in Overweight/Obese Patients With Newly Diagnosed Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Director of Endocrinology,Principal Investigator, Beijing Chao Yang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-科 144
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Exenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exenatide group (Experimental): The drug-naïve, overweight or obese patients with newly diagnosed T2D
  Interventions: Drug: Exenatide or metformin hydrochloride
- metformin group (Active Comparator): The drug-naïve, overweight or obese patients with newly diagnosed T2D
  Interventions: Drug: Exenatide or metformin hydrochloride

INTERVENTIONS:
Drug: Exenatide or metformin hydrochloride — Exenatide was administrated with 5 μg bid for 4 weeks and 10 μg bid for 8 weeks. Metformin hydrochloride was initiated at a dose of 500 mg bid for 2 weeks, and added to 2.0 g/day for 8 weeks.

SUMMARY:
The present study assessed the therapeutic effect of exenatide and metformin as the initial therapy in overweight/obese patients with newly diagnosed Type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The present study was a prospective, nonrandomized, interventional study.The drug-naïve, overweight or obese patients with newly diagnosed T2D were consecutively enrolled. The inclusion criteria: 1) age 20 - <65 years, 2) body mass index (BMI) ≥ 24 kg/m2 [7], and 3) HbA1c ≥ 7% (53mmol/mol). An oral glucose tolerance test was performed during the screenings. All of the patients have no diabetes antibodies and were diagnosed with T2D within the previous 3 months, according to the ADA diagnostic criteria. None of the patients had administered anti-diabetic drugs or diet therapy before participation. Neither of the patients presented any history of pancreatitis, coronary artery disease, liver function impairment, renal function impairment, intestinal surgery, chronic hypoxic diseases (emphysema and cor pulmonale), infectious disease, hematological disease, systemic inflammatory disease, or cancer. Patients who were pregnant, possibly pregnant, or ingesting agents known to influence glucose or lipid metabolism were also excluded.

ELIGIBILITY:
Inclusion Criteria:

* age 20 - <65 years,
* body mass index (BMI) ≥ 24 kg/m2,
* HbA1c ≥ 7% (53mmol/mol).
* diabetes antibodies (-)
* diagnosed with T2D within the previous 3 months

Exclusion Criteria:

* anti-diabetic drugs or diet therapy before participation
* pancreatitis
* coronary artery disease
* liver function impairment
* renal function impairment
* intestinal surgery
* chronic hypoxic diseases (emphysema and cor pulmonale)
* infectious disease
* hematological disease
* systemic inflammatory disease
* cancer
* pregnant, possibly pregnant
* ingesting agents known to influence glucose or lipid metabolism

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
The change of HbA1c | baseline and 12 weeks

REFERENCES:
- [Derived] Zhang L, Hu Y, An Y, Wang Q, Liu J, Wang G. The Changes of Lipidomic Profiles Reveal Therapeutic Effects of Exenatide in Patients With Type 2 Diabetes. Front Endocrinol (Lausanne). 2022 Mar 31;13:677202. doi: 10.3389/fendo.2022.677202. eCollection 2022. PMID 35432194
- [Derived] Liu J, Hu Y, Xu Y, Jia Y, Miao L, Wang G. Comparison of Exenatide and Metformin Monotherapy in Overweight/Obese Patients with Newly Diagnosed Type 2 Diabetes. Int J Endocrinol. 2017;2017:9401606. doi: 10.1155/2017/9401606. Epub 2017 Nov 20. PMID 29358950